CLINICAL TRIAL: NCT05292950
Title: A Phase 1/2a Study Evaluating the Effects of ARO-MUC5AC Inhalation Solution in Healthy Subjects and Patients With Muco-Obstructive Lung Disease
Brief Title: Study of ARO-MUC5AC in Healthy Subjects and Patients With Muco-Obstructive Lung Disease
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Sponsor business decision
Sponsor: Arrowhead Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: AROMUC5AC-1001; 2022-003467-21 (EudraCT Number)
Record Dates: First submitted 2022-03-15; First posted 2022-03-23 (Actual); Last update posted 2025-11-05 (Actual); Status verified 2025-11

CONDITIONS: Asthma; Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Asthma; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- ARO-MUC5AC (Experimental): ARO-MUC5AC Inhalation
  Interventions: Drug: ARO-MUC5AC
- Placebo (Placebo Comparator): (0.9% NaCl)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ARO-MUC5AC — single or multiple doses of ARO- MUC5AC by inhalation of nebulized solution
  Arms: ARO-MUC5AC
Drug: Placebo — calculated volume to match active treatment by inhalation of nebulized solution
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, and pharmacokinetics (PK) of ARO-MUC5AC in normal healthy volunteers (NHVs), patients with moderate-to-severe asthma and patients with moderate-to-severe chronic obstructive pulmonary disease (COPD). In part 1 NHVs will receive a single dose of ARO-MUC5AC or placebo. In part 2 of the study, NHVs, adult patients with asthma, and adult patients with COPD will receive 3 doses of ARO-MUC5AC or placebo.

ELIGIBILITY:
Inclusion Criteria:

* Normal pulmonary function tests at Screening (NHVs only)
* Confirmed diagnosis of asthma or COPD based on source verifiable medical record (asthma and COPD patients only)
* No abnormal finding of clinical relevance at Screening (NHVs only)
* Stable dose of asthma controller medications for at least 28 days prior to Screening (asthma patients only)
* Documented treatment with an inhaled corticosteroid and at least 1 additional maintenance asthma controller medication for at least 3 months prior to Screening (asthma patients only)
* Non-smoking (NHVs and asthma patients)
* Current smoker or ex-smoker with smoking history of ≥ 10 pack-years (COPD patients only)
* All COPD treatments have been stable for at least one month prior to Screening (COPD patients only)
* Able to produce an induced sputum sample at Screening
* Women of childbearing potential must have a negative pregnancy test, cannot be breastfeeding, and must be willing to use contraception. Males must not donate sperm during the study and for at least 90 days following the last dose of study drug
* Willing to provide written informed consent and to comply with study requirements

Exclusion Criteria:

* Acute lower respiratory infection within 30 days prior to first dose and/or acute upper respiratory infection within 7 days prior to first dose
* Positive COVID-19 test during Screening window
* Any history of chronic pulmonary disease (NHVs only)
* Any concomitant pulmonary disease in asthma or COPD patients that could interfere with the evaluation of the study drug or interpretation of patient safety or study results
* Use of theophylline within 30 days prior to first dose
* History of lung volume reduction surgery or pneumonectomy (COPD patients)
* Need for chronic oxygen support at Screening
* Clinically significant health concerns (other than asthma in asthma patients)
* Human immunodeficiency virus (HIV) infection, seropositive for hepatitis B virus (HBV), seropositive for hepatitis C virus (HCV)
* Uncontrolled hypertension
* Unwilling to limit alcohol consumption to within moderate limits for the duration of the study
* Use of illicit drugs
* Use of an investigational agent or device within 30 days prior to first dose

Note: additional inclusion/exclusion criteria may apply per protocol

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2022-06-27 (Actual); Primary Completion 2024-11-12 (Actual); Study Completion 2024-11-12 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Treatment-Emergent Adverse Events (TEAEs) | single dose phase: up to Day 29; multiple dose phase: up to Day 85

SECONDARY OUTCOMES:
Change Over Time from Baseline in Forced Expiratory Volume (FEV1) | single dose phase: up to Day 29; multiple dose phase: up to Day 85
Change Over Time from Baseline in Forced Vital Capacity (FVC) | single dose phase: up to Day 29; multiple dose phase: up to Day 85
PK of ARO-MUC5AC: Maximum Observed Plasma Concentration (Cmax) | single dose phase: up to 48 Hours; multiple dose phase: up to 6 hours post-dose on Days 1 and 29 for NHVs; and up to 6 hours post-dose on Days 1 and 29, and up to 24 hours post-dose on Days 2 and 30 for participants with asthma or COPD
PK of ARO-MUC5AC: Area Under the Plasma Concentration versus Time Curve From Zero to 24 Hours (AUC0-24) | single dose phase: up to 48 Hours; multiple dose phase: up to 6 hours post-dose on Days 1 and 29 for NHVs; and up to 6 hours post-dose on Days 1 and 29, and up to 24 hours post-dose on Days 2 and 30 for participants with asthma or COPD
PK of ARO-MUC5AC: Area Under the Plasma Concentration versus Time Curve From Zero to the Last Quantifiable Plasma Concentration (AUClast) | single dose phase: up to 48 Hours; multiple dose phase: up to 6 hours post-dose on Days 1 and 29 for NHVs; and up to 6 hours post-dose on Days 1 and 29, and up to 24 hours post-dose on Days 2 and 30 for participants with asthma or COPD
PK of ARO-MUC5AC: Area Under the Plasma Concentration versus Time Curve From Zero to Infinity (AUCinf) | single dose phase: up to 48 Hours; multiple dose phase: up to 6 hours post-dose on Days 1 and 29 for NHVs; and up to 6 hours post-dose on Days 1 and 29, and up to 24 hours post-dose on Days 2 and 30 for participants with asthma or COPD
PK of ARO-MUC5AC: Terminal Elimination Half-Life (t1/2) | single dose phase: up to 48 Hours; multiple dose phase: up to 6 hours post-dose on Days 1 and 29 for NHVs; and up to 6 hours post-dose on Days 1 and 29, and up to 24 hours post-dose on Days 2 and 30 for participants with asthma or COPD
PK of ARO-MUC5AC: Apparent Systemic Clearance (CL/F) | single dose phase: up to 48 Hours; multiple dose phase: up to 6 hours post-dose on Days 1 and 29 for NHVs; and up to 6 hours post-dose on Days 1 and 29, and up to 24 hours post-dose on Days 2 and 30 for participants with asthma or COPD
PK of ARO-MUC5AC: Apparent Terminal-Phase Volume of Distribution (VZ/F) | single dose phase: up to 48 Hours; multiple dose phase: up to 6 hours post-dose on Days 1 and 29 for NHVs; and up to 6 hours post-dose on Days 1 and 29, and up to 24 hours post-dose on Days 2 and 30 for participants with asthma or COPD
PK of ARO-MUC5AC: Recovery of Unchanged Drug in Urine Over 24 Hours (Amount Excreted; Ae) | through 24 hours post-dose
PK of ARO-MUC5AC: Percentage of Administered Drug Recovered in Urine Over 0-24 Hours | through 24 hours post-dose
PK of ARO-MUC5AC: Renal Clearance (CLr) | single dose phase: up to 48 Hours; multiple dose phase: up to 6 hours post-dose on Days 1 and 29 for NHVs; and up to 6 hours post-dose on Days 1 and 29, and up to 24 hours post-dose on Days 2 and 30 for participants with asthma or COPD

CONTACTS AND LOCATIONS:
Locations (13):
- Australia (2):
  - Research Site 2, South Brisbane, Queensland
  - Research Site 1, Nedlands
- New Zealand (2):
  - Research Site 1, Auckland
  - Research Site 2, Auckland
- Poland (3):
  - Research Site 1, Bialystok
  - Research Site 2, Krakow
  - Research Site 3, Oświęcim
- South Korea (3):
  - Research Site 3, Bucheon-si, Gyeonggi-do
  - Research Site 2, Jeonju
  - Research Site 1, Seoul
- Research Site 1, Barcelona, Spain
- Research Site 1, Bangkok, Thailand
- Research Site 1, Wythenshawe, Manchester, United Kingdom